CLINICAL TRIAL: NCT03020992
Title: Multicenter, Open-Label Study to Assess the Effects of Certolizumab Pegol on the Reduction of Anterior Uveitis Flares in Axial Spondyloarthritis Subjects With a History of Anterior Uveitis (C-VIEW)
Brief Title: A Study to Assess the Effects of Certolizumab Pegol on the Reduction of Anterior Uveitis (AU) Flares in Axial Spondyloarthritis Subjects With a Documented History of AU
Acronym: C-VIEW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS0007; 2016-000343-14 (EudraCT Number)
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Axial Spondyloarthritis (axSpA); Anterior Uveitis (AU)
Keywords: Axial Spondyloarthritis; axSpA; Anterior Uveitis; Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Axial Spondyloarthritis; Uveitis, Anterior | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Certolizumab Pegol (Experimental): Subjects will receive a loading dose of Certolizumab Pegol (CZP) 400 mg subcutaneously (sc) administered at Baseline, Week 2, and Week 4 followed by CZP 200 mg sc every two Weeks
  Interventions: Drug: Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol — * pharmaceutical form: solution for infusion in prefilled syringe
  * concentration: 200 mg/mL
  * route of administration: subcutaneous
  Other Names: Cimzia; CZP; CDP870

SUMMARY:
The purpose of the study is to demonstrate the effect of Certolizumab Pegol (CZP) treatment on the reduction of Anterior Uveitis (AU) flares in subjects with active axial Spondyloarthritis (axSpA) and a documented history of AU.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a documented diagnosis of adult-onset axial Spondyloarthritis (axSpA) with at least 3 months' symptom duration and meet the Assessment of SpondyloArthritis International Society (ASAS) criteria
* Subjects must have active disease at Screening as defined by
* Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score >= 4
* Spinal pain >= 4 on a 0 to 10 Numerical Rating Scale (NRS; from BASDAI item 2)
* Nonradiographic (Nr)-axSpA subjects must either have C-reactive protein (CRP) > upper limit of normal (ULN) and /or current evidence of sacroiliitis on magnetic resonance imaging (MRI) (no confirmation by central reading) as defined by ASAS criteria
* Ankylosing spondylitis (AS) subjects must have evidence of sacroiliitis on x-ray meeting the modified New York (mNY) classification criteria according to the Investigator
* Subjects must have a documented history of Anterior Uveitis (AU) diagnosed by an ophthalmologist and have at least 2 AU flares in the past, of which at least 1 AU flare was in the last 12 months prior to Baseline

Exclusion Criteria:

* Other inflammatory arthritis
* Secondary, noninflammatory condition that, in the Investigator's opinion, is symptomatic enough to interfere with evaluation of the effect of study drug on the subject's primary diagnosis of axial spondyloarthritis (axSpA)
* Any history of uveitis except for Anterior Uveitis (AU) associated with axSpA
* Any condition or complicating factor that may interfere with the AU assessment
* Retisert® or Iluvien® (glucocorticosteroid implant) within 3 years prior to the Baseline Visit or has had complications related to the device
* Subject has had Retisert or Iluvien (glucocorticosteroid implant) removed within 90 days prior to the Baseline Visit
* Intraocular or periocular corticosteroids within 90 days prior to the Baseline visit
* Ozurdex® (dexamethasone implant) within 6 months prior to the Baseline Visit
* Cyclophosphamide within 30 days prior to the Baseline Visit
* Intravitreal methotrexate (MTX) within 90 days prior to the Baseline Visit
* Intravitreal anti-vascular endothelial growth factor (VEGF) therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2020-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (23):
- Czechia (7):
  - As0007 101, Brno
  - As0007 103, Brno
  - As0007 107, Brno
  - As0007 108, Ostrava
  - As0007 109, Pardubice
  - As0007 102, Prague
  - As0007 105, Prague
- Germany (3):
  - As0007 301, Freiburg im Breisgau
  - As0007 302, München
  - As0007 303, Münster
- As0007 401, Amsterdam, Netherlands
- Poland (10):
  - As0007 506, Bialystok
  - As0007 510, Lublin
  - As0007 509, Poznan
  - As0007 511, Poznan
  - As0007 502, Torun
  - As0007 501, Warsaw
  - As0007 505, Warsaw
  - As0007 504, Wroclaw
  - As0007 507, Wroclaw
  - As0007 508, Wroclaw
- Spain (2):
  - As0007 604, Barcelona
  - As0007 601, Córdoba

REFERENCES:
- [Derived] van der Horst-Bruinsma IE, van Bentum RE, Verbraak FD, Deodhar A, Rath T, Hoepken B, Irvin-Sellers O, Thomas K, Bauer L, Rudwaleit M. Reduction of anterior uveitis flares in patients with axial spondyloarthritis on certolizumab pegol treatment: final 2-year results from the multicenter phase IV C-VIEW study. Ther Adv Musculoskelet Dis. 2021 Mar 29;13:1759720X211003803. doi: 10.1177/1759720X211003803. eCollection 2021. PMID 33854572
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled in December 2016 and the last participant was enrolled in December 2017.
Pre-assignment Details: The study included 3 periods as follows: Period 1 (Screening Period) 1 to 5 weeks before Baseline, Period 2 (Treatment Period) Week 0 to Week 96 and Period 3 (FU Period) 10 weeks from the final dose of investigational medicinal product (IMP) received (Week 104).
  Participant Flow refers to the Safety Set.
Groups:
- Certolizumab Pegol: Participants received a loading dose of Certolizumab Pegol (CZP) 400 milligrams (mg) subcutaneously (sc) administered at Baseline, Week 2, and Week 4 followed by CZP 200 mg sc every 2 weeks (Q2W) (starting at Week 6 until Week 94).
Period: Overall Study
Arm/Group | Certolizumab Pegol
Started | 89
Completed | 83
Not Completed | 6
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The Safety Set (SS) consisted of all study participants in the Enrolled Set (ES) who had received at least 1 dose of IMP.
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 84
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.52 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87
  Other or Mixed | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Distinct Episodes of Anterior Uveitis (AU) Flares During the Treatment Period
Description: A flare was defined as being a new episode of Anterior Uveitis (AU) that, based on the judgment of an ophthalmologist, required specific treatment. A flare was considered a new episode if a gap of at least 3 months occurred between 2 flares.
Time Frame: During the pre-study period and during the Treatment Period up to 96 weeks
Population: The Full Analysis Set (FAS) consisted of all study participants in the Safety Set (SS) with nonmissing Baseline values for the primary efficacy variable (AU flare incidence data from the prestudy period).
Measure: Mean (Standard Deviation); unit: flares
Groups:
- Certolizumab Pegol (FAS): Participants received a loading dose of Certolizumab Pegol (CZP) 400 mg subcutaneously (sc) administered at Baseline, Week 2, and Week 4 followed by CZP 200 mg sc Q2W (starting at Week 6 until Week 94).
Arm/Group | Certolizumab Pegol (FAS)
Number analyzed (Participants) | 89
flares
  Pre-study Historical | 1.9 (0.9)
  On-study CZP | 0.3 (0.7)
Statistical Analysis 1: Comparison: Certolizumab Pegol (FAS); The Poisson regression allowed for a comparison of event rates adjusting for differences in time between prestudy/on-study periods. Event rates were based on a Poisson model with generalized estimating equations and a log-link, including an offset term for time interval length, and with period and disease duration of axSpA (<2 years/≥2 years) as covariates. A repeated statement was included for participants and assumed an exchangeable correlation structure between prestudy and on-study flares; Test type: Other; p < 0.001, Poisson regression; Rate ratio = 0.180, 95% CI 2-sided [0.116 to 0.281]

2. Secondary Outcome: Number of Anterior Uveitis (AU) Flares Per 100 Patient-years in Participants With Active Axial SpondyloArthritis (axSpA) and a History of AU at Week 48
Description: as for outcome 1
Time Frame: During the pre-study period and during the Treatment Period up to 48 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: flares
Arm/Group | Certolizumab Pegol (FAS)
Number analyzed (Participants) | 89
flares
  Pre-study Historical | 132.72 [109.76 to 159.06]
  On-study CZP | 18.56 [10.39 to 30.61]

3. Secondary Outcome: Number of Anterior Uveitis (AU) Flares Per 100 Patient-years in Participants With Active Axial SpondyloArthritis (axSpA) and a History of AU at Week 96
Description: as for outcome 1
Time Frame: During the pre-study period and during the Treatment Period up to 96 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: flares
Arm/Group | Certolizumab Pegol (FAS)
Number analyzed (Participants) | 89
flares
  Pre-study Historical | 97.51 [83.24 to 113.53]
  On-study CZP | 17.67 [11.74 to 25.53]

4. Secondary Outcome: Number of Anterior Uveitis (AU) Flares Per 100 Patient-years in Participants With Active Axial SpondyloArthritis (axSpA) and at Least 1 AU Episode Within 12 Months Prior Baseline at Week 48
Description: as for outcome 1
Time Frame: During the pre-study period and during the Treatment Period up to 48 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: flares
Arm/Group | Certolizumab Pegol (FAS)
Number analyzed (Participants) | 89
flares
  Pre-study Historical | 132.72 [109.76 to 159.06]
  On-study CZP | 18.56 [10.39 to 30.61]

5. Secondary Outcome: Number of Anterior Uveitis (AU) Flares Per 100 Patient-years in Participants With Active Axial SpondyloArthritis (axSpA) and at Least 1 AU Episode Within 12 Months Prior Baseline at Week 96
Description: as for outcome 1
Time Frame: During the pre-study period and during the Treatment Period up to 96 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: flares
Arm/Group | Certolizumab Pegol (FAS)
Number analyzed (Participants) | 89
flares
  Pre-study Historical | 97.51 [83.24 to 113.53]
  On-study CZP | 17.67 [11.74 to 25.53]

6. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 48
Description: The ASDAS was calculated as the sum of the following:
  0.121 × Back pain (Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Question 2 result) 0.058 × Duration of morning stiffness (BASDAI Question 6 result) 0.110 × Patient's Global Assessment of Disease Activity (PtGADA) 0.073 × Peripheral pain/swelling (BASDAI Question 3 result) 0.579 × (natural logarithm (C-Reactive Protein (CRP) [mg/L] + 1)) Back pain, PtGADA, duration of morning stiffness, and peripheral pain/swelling are all assessed on a numerical scale (0 to 10 units).
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
  There is a minimum score of 0.636 for the total ASDAS score, but no defined upper score. Based on the formula even in the situation that the CRP is normal, any value below 4 is recorded as 'below the limit of quantification' (BLQ) and a value of BLQ/2=2 was prespecified. This assumption is triggering the lowest possible value of 0.636.
Time Frame: From Baseline to Week 48
Population: The Safety Set consisted of all study participants in the Enrolled Set (ES) who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing ASDAS at Week 48.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Certolizumab Pegol (SS): Participants received a loading dose of Certolizumab Pegol (CZP) 400 mg subcutaneously (sc) administered at Baseline, Week 2, and Week 4 followed by CZP 200 mg sc Q2W (starting at Week 6 until Week 94).
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 86
scores on a scale | -1.55 (1.03)

7. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 96
Description: as for outcome 6
Time Frame: From Baseline to Week 96
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing ASDAS at Week 96.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 82
scores on a scale | -1.61 (1.08)

8. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 48
Description: The BASDAI is a validated self-reported instrument which consists of 6 horizontal Numeric Rating Scales (NRSs), each with 10 units to measure the severity of the 5 major symptoms: fatigue, spinal pain, peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. To give each symptom equal weighting, the average of the 2 scores relating to morning stiffness is taken. The resulting 0 to 50 sum score is divided by 5 to give a final BASDAI score between 0 and 10, with lower scores indicating lower disease activity.
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 48
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing BASDAI at Week 48.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 86
scores on a scale | -3.2 (2.3)

9. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 96
Description: as for outcome 8
Time Frame: From Baseline to Week 96
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing BASDAI at Week 96.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 82
scores on a scale | -3.4 (2.2)

10. Secondary Outcome: Percentage of Participants Meeting Assessment of SpondyloArthritis International Society 20 % Response Criteria (ASAS20) at Week 48
Description: The ASAS20 is defined as an improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 following domains and absence of deterioration in the potential remaining domain [deterioration was defined as a relative worsening of at least 20 % and an absolute worsening of at least 1 unit]:
  * Patient's Global Assessment of Disease Activity (PtGADA)
  * Pain assessment (the total spinal pain Numeric Rating Scale score)
  * Function (represented by Bath Ankylosing Spondylitis Functional Index (BASFI))
  * Inflammation (the mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration)
Time Frame: Week 48
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Percentages were based on the number of participants with an assessment at Week 48.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 86
percentage of participants | 75.6

11. Secondary Outcome: Percentage of Participants Meeting Assessment of SpondyloArthritis International Society 20 % Response Criteria (ASAS20) at Week 96
Description: as for outcome 10
Time Frame: Week 96
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Percentages were based on the number of participants with an assessment at Week 96.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 82
percentage of participants | 75.6

12. Secondary Outcome: Percentage of Participants Meeting Assessment of SpondyloArthritis International Society 40 % Response Criteria (ASAS40) at Week 48
Description: The ASAS criteria for 40 % improvement were defined as relative improvements of at least 40 %, and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains below and no worsening at all in the remaining domain:
  * Patient's Global Assessment of Disease Activity (PtGADA)
  * Pain assessment (the total spinal pain Numeric Rating Scale score)
  * Function (represented by Bath Ankylosing Spondylitis Functional Index (BASFI))
  * Inflammation (the mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration)
Time Frame: Week 48
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 86
percentage of participants | 53.5

13. Secondary Outcome: Percentage of Participants Meeting Assessment of SpondyloArthritis International Society 40 % Response Criteria (ASAS40) at Week 96
Description: as for outcome 12
Time Frame: Week 96
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 82
percentage of participants | 58.5

14. Secondary Outcome: Percentage of Participants Meeting Assessment of SpondyloArthritis International Society (ASAS) 5/6 Response at Week 48
Description: The ASAS 5/6 response is defined as at least 20 % improvement in 5 of 6 domains, including spinal mobility (lateral spinal flexion) and C-Reactive Protein (CRP) as more objective measures.
  As the BASMI was not collected, and there was no alternative measure of spinal mobility available in the study data, the complete component for spinal mobility was missing. Therefore the ASAS 5/6 response criterion cannot be calculated, and the analysis of the secondary efficacy variable ASAS 5/6 had to be dropped.
Time Frame: Week 48
Population: Data not collected from participants in all Arms/Groups.
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 0

15. Secondary Outcome: Percentage of Participants Meeting Assessment of SpondyloArthritis International Society (ASAS) 5/6 Response at Week 96
Description: as for outcome 14
Time Frame: Week 96
Population: Data not collected from participants in all Arms/Groups.
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 0

16. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society (ASAS) Partial Remission (PR) Response at Week 48
Description: The ASAS PR response is defined as a score of ≤2 units on a 0 to 10 unit scale in all of the 4 following domains:
  * Patient's Global Assessment of Disease Activity (PtGADA)
  * Pain assessment (the total spinal pain Numeric Rating Scale score)
  * Function (represented by Bath Ankylosing Spondylitis Functional Index (BASFI))
  * Inflammation (the mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration)
Time Frame: Week 48
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 86
percentage of participants | 31.4

17. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society (ASAS) Partial Remission (PR) Response at Week 96
Description: as for outcome 16
Time Frame: Week 96
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 82
percentage of participants | 36.6

18. Secondary Outcome: Change From Baseline in Tender Joint Count (44 Joint Count) at Week 48
Description: The following 44 joints were to be examined for swelling and tenderness by the Investigator, another delegated physician, or an appropriately qualified medical professional:
  * Upper body (4) - bilateral sternoclavicular and acromioclavicular joints
  * Upper extremity (26) - bilateral shoulders, elbows, wrists (includes radiocarpal, carpal, and carpometacarpal bones considered as a single unit), metacarpophalangeals (MCPs) I,II, III, IV, and V, and thumb interphalangeals (IPs), and proximal IPs (PIPs) II, III, IV, and V
  * Lower extremity (14) - bilateral knees, ankles, and metatarsophalangeals (I, II, III, IV, and V) The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 48
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with at least one tender joint count at Baseline (N=59) and had a non-missing tender joint count at Week 48 (N=55).
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 55
tender joints | -4.9 (6.7)

19. Secondary Outcome: Change From Baseline in Tender Joint Count (44 Joint Count) at Week 96
Description: as for outcome 18
Time Frame: From Baseline to Week 96
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with at least one tender joint count at Baseline (N=59) and had a non-missing tender joint count at Week 96 (N=51).
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 51
tender joints | -4.7 (8.2)

20. Secondary Outcome: Change From Baseline in Swollen Joint Count (44 Joint Count) at Week 48
Description: as for outcome 18
Time Frame: From Baseline to Week 48
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with at least one swollen joint count at Baseline (N=33) and had a non-missing swollen joint count at Week 48 (N=32).
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 32
swollen joints | -4.2 (4.8)

21. Secondary Outcome: Change From Baseline in Swollen Joint Count (44 Joint Count) at Week 96
Description: as for outcome 18
Time Frame: From Baseline to Week 96
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with at least one swollen joint count at Baseline (N=33) and had a non-missing swollen joint count at Week 96 (N=30).
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 30
swollen joints | -3.9 (5.2)

22. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity (PhGADA) at Week 48
Description: The Investigator assessed the overall status of the participant with respect to the axSpA signs and symptoms and the functional capacity of the participant using a Visual Analog Scale (VAS) where 0 is "very good, asymptomatic and no limitation of normal activities" and 100 is "very poor, very severe symptoms that are intolerable, and the inability to carry out all normal activities." This assessment by the Investigator should be made without any knowledge of the Patient's Global Assessment of Disease Activity (PtGADA).
  Total score ranges from 0 to 100, with lower scores indicating lower disease activity.
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 48
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing PhGADA at Week 48.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 86
scores on a scale | -43.8 (21.6)

23. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity (PhGADA) at Week 96
Description: as for outcome 22
Time Frame: From Baseline to Week 96
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing PhGADA at Week 96.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 82
scores on a scale | -42.5 (27.1)

24. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity (PtGADA) at Week 48
Description: For the PtGADA questionnaire, participants scored their global assessment of their disease activity in response to the question "How active was your spondylitis on average during the last week?" using a Numeric Rating Scale (NRS) where 0 was "not active" and 10 was "very active".
  Total score ranges from 0 to 10, with lower scores indicating lower disease activity.
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 48
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing PtGADA at Week 48.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 86
scores on a scale | -3.6 (2.5)

25. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity (PtGADA) at Week 96
Description: as for outcome 24
Time Frame: From Baseline to Week 96
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing PtGADA at Week 96.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 82
scores on a scale | -3.9 (2.7)

26. Secondary Outcome: Change From Baseline in Total Spinal Pain at Week 48 Assessed by Numerical Rating Scale (NRS)
Description: The total spinal pain was assessed with the question 'How much pain of your spine due to spondylitis do you have?' using a Numeric Rating Scale (NRS) where 0 was 'No pain' and 10 was 'Most severe pain'. Usually, a 10 % difference (ie, a 1 point difference on a Numeric Rating Scale (NRS) ranging from 0 to 10) is considered the minimal clinically important difference used to interpret scores (Dworkin et al, 2008).
  Total score ranges from 0 to 10, with lower scores indicating a worse outcome. The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 48
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing total spinal pain assessment at Week 48.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 86
scores on a scale | -3.8 (2.5)

27. Secondary Outcome: Change From Baseline in Total Spinal Pain at Week 96 Assessed by Numerical Rating Scale (NRS)
Description: as for outcome 26
Time Frame: From Baseline to Week 96
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing total spinal pain assessment at Week 96.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 82
scores on a scale | -4.1 (2.6)

28. Secondary Outcome: Change From Baseline to Week 48 in the Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The BASFI is a validated disease-specific instrument for assessing physical function (van Tubergen et al, 2015; Calin et al, 1994; van der Heijde et al, 2005).
  The BASFI comprises 10 items relating to the past week. The Numeric Rating Scale (NRS) version was used for the answering options of each item on a scale of 0 ("Easy") to 10 ("Impossible") (van Tubergen et al, 2002). The BASFI score is the mean of the 10 items such that the total score ranges from 0 to 10, with lower scores indicating better physical function.
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 48
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing BASFI at Week 48.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 86
scores on a scale | -2.23 (2.33)

29. Secondary Outcome: Change From Baseline to Week 96 in the Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: as for outcome 28
Time Frame: From Baseline to Week 96
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
  Number of participants analyzed reflect those with a non-missing BASFI at Week 96.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 82
scores on a scale | -2.28 (2.53)

30. Secondary Outcome: Change From Baseline to Week 48 in Inflammation Assessed by the Mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Questions 5 and 6 Concerning Morning Stiffness and Duration
Description: The BASDAI is a validated self-reported instrument which consists of six 10-unit horizontal Numeric Rating Scales (NRS) to measure severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration for each disease activity, respectively) over the last week. The mean of the 2 BASDAI questions related to morning stiffness (questions 5 and 6) ranged from 0 to 10, with lower scores indicating lower disease activity.
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 86
scores on a scale | -3.7 (2.8)

31. Secondary Outcome: Change From Baseline to Week 96 in Inflammation Assessed by the Mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Questions 5 and 6 Concerning Morning Stiffness and Duration
Description: as for outcome 30
Time Frame: From Baseline to Week 96
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 82
scores on a scale | -3.8 (2.7)

32. Secondary Outcome: Percentage of Participants Reporting at Least One Treatment-Emergent Adverse Events (TEAEs) During the Study
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Baseline up to the Safety Follow-up Visit (up to Week 104)
Population: The Safety Set consisted of all study participants in the Enrolled Set who had received at least 1 dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol (SS)
Number analyzed (Participants) | 89
percentage of participants | 80.9

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from Baseline to the Safety Follow-up Visit (up to Week 104)
Arm/Group | Certolizumab Pegol (SS)
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 11/89
Other Adverse Events (participants affected / at risk) | 51/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (SS) (N=89)
Vestibular disorder (Ear and labyrinth disorders) | 2 (2)
Uveitis (Eye disorders) | 1 (2)
Anal polyp (Gastrointestinal disorders) | 1 (1)
Incarcerated hernia (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (SS) (N=89)
Uveitis (Eye disorders) | 14 (23)
Iridocyclitis (Eye disorders) | 8 (12)
Nasopharyngitis (Infections and infestations) | 15 (22)
Upper respiratory tract infection (Infections and infestations) | 12 (15)
Influenza (Infections and infestations) | 6 (9)
Rhinitis (Infections and infestations) | 6 (9)
Alanine aminotransferase increased (Investigations) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT03020992/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03020992/SAP_001.pdf